CLINICAL TRIAL: NCT06927635
Title: Stereotactic Body Radiotherapy or Standard of Care for Prostate Oligoprogressive Cancer: a Randomized Phase II Trial
Brief Title: Stereotactic Body Radiotherapy or Standard of Care for Prostate Oligoprogressive Cancer
Acronym: SECURE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-5872
Record Dates: First submitted 2025-03-03; First posted 2025-04-15 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Castrate Resistance Prostate Cancer; OligoProgressive Metastatic Disease
Keywords: systemic therapy; stereotactic body radiation therapy (SBRT)
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 - Standard of Care (Active Comparator): Participants on Arm 1 - SOC will be treated as per standard of care by their treating Oncologist. In most instances, it is anticipated participants will undergo a change in Systemic Therapy (ST) (including best supportive care). The ST will be at the discretion of the Oncologist and patient, according to best practices for the patient's diagnosis and clinical scenario. Patients can receive palliative radiotherapy for standard indications at any time.
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT); Other: Systemic therapy
- Arm 2 - Experimental (Experimental): Participants on Arm 2 - Experimental will receive standard of care SBRT to oligoprogressive sites according to institutional standards while remaining on the systemic treatment prescribed by the treating oncologist.
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT); Other: Systemic therapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) — SBRT will be delivered as per institutional standard.
Other: Systemic therapy — Participants will receive Systemic Therapy. Participants in Arm 1 - SOC may change the Systemic Therapy throughout treatment. Participants in Arm 2 - Experimental will remain on the same Systemic Therapy throughout treatment.

SUMMARY:
This is a single centre, interventional, randomized Phase II, two-arm prospective trial investigating if Stereotactic Body Radiotherapy (SBRT) to all sites of Oligopressive (OP) disease while remaining on current Systemic Therapy (ST) will improve biochemical control compared to Standard of Care (SoC) (which involves a change in ST) for patients with OP Castrate Resistance Prostate Cancer (CRPC).

DETAILED DESCRIPTION:
The current standard of care for patients with metastatic Oligopressive (OP) Castrate Resistance Prostate Cancer (CRPC) is a change in Systemic Therapy (ST). We propose that Stereotactic Body Radiotherapy (SBRT) to Oligopressive sites, while maintaining patients on their current Systemic Therapy, may allow for biochemical control of disease while maintaining patient Quality of Life and avoiding the toxicities associated with changing Systemic Therapy. We have proposed an initial prospective feasibility study, followed by a larger phase II prospective study to investigate the efficacy of SBRT in Oligopressive Castrate Resistance Prostate Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Able to provide informed consent
* Histologic diagnosis of prostate adenocarcinoma
* Castrate Resistance Prostate Cancer
* Radiographic evidence of <10 sites of extra-cranial OP metastatic lesions
* Receiving any line of ST for >3 months
* All sites of OP disease are amenable to and can be safely treated with SBRT
* ECOG performance status 0-3

Exclusion Criteria:

* Evidence of spinal cord compression
* Contraindication to radiotherapy

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must be male due to the disease site (prostate).
Enrollment: 75 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Study Feasibility | Within 18 months of study activation.
  Determine the feasibility of enrolling 21 patients patients onto a study randomizing patients to either MDT using SBRT plus remaining on current ST versus SoC (change in Systemic Therapy) by measuring the rate accrual (number of patients per month for 18 months).
Change in Prostate-Specific Antigen (PSA) | Enrollment to 12 months post-enrollment.
  Assess by standard PSA blood testing if the proportion of patients having a >50% change in PSA compared to baseline (PSA50) is improved with MDT using SBRT plus remaining on current ST versus SoC.

SECONDARY OUTCOMES:
Radiographic Local Control of Oligopressive Lesions | Enrollment to 12 months-post enrollment.
  Radiographic local control of the index OP lesions will be assessed by treating oncologist.
Radiographic Distant Control of Oligopressive Lesions | Enrollment to 12-months post-enrollment.
  Defined by growth of non-Oligoprogressive metastatic sites and/or the development of new sites of metastatic disease, as assessed by treating oncologist.
Progression Free Survival (PFS) | Enrollment to 12-months post-enrollment.
  Defined as the time from randomization to death from any cause, progression of disease, or date of last follow-up, whichever occurs first. PFS will be assessed by the treating oncologist.
Time to next Systemic Therapy | Enrollment to 12-months post-enrollment.
  Defined as the time from when the study intervention has been commenced until commencement of any next systemic anti-cancer therapy (including a change to best supportive care) or date of last follow up, whichever occurs first, which will be assess by the treating oncologist.
Differences in Toxicity | Enrollment to 12-months post-enrollment.
  Toxicity will be assessed to determine whether SBRT compared to SoC results in patient- and/or physician-reported toxicity differences. Toxicity will be collected using CTCAE v5.0
Differences in Quality of Life | Enrollment to 12-months post-enrollment.
  Quality of Life (QoL) will be assessed to determine whether SBRT compared to SoC results in patient- and/or physician-reported QoL differences. QoL will be collected using the EORTC QLQ-C30 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Glicksman, MD, Principal Investigator — Princess Margaret Cancer Centre - University Health Network
Locations (1):
- Princess Margaret Cancer Center, Toronto, Ontario, Canada